CLINICAL TRIAL: NCT06631339
Title: Optimizing Light Exposure for Myopia Prevention and Control (LightSPAN)
Acronym: LightSPAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Technical University of Munich Campus for Research Excellence And Technological Enterprise (TUMCREATE) (Unknown)
Responsible Party: Principal Investigator, Raymond P. Najjar, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-767
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Light; Therapy, Complications; Myopia Progression; Short-Sighted; Myopia; Refractive Error
Keywords: Light Exposure; Digital Intervention; Myopia; Myopia Prevention; Cognition; Light Intervention; Behaviour changing phone application; Classroom; School-based; School; Singapore; Primary School; Light therapy; Myopia-control
MeSH Terms: conditions — Myopia; Refractive Errors | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Primary School-based, 12-Month, semi-randomised, controlled, double-blinded, 3 study arm (n=132 per arm) trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind, semi-randomised controlled trial in which neither the study participants, the investigators nor study personnel responsible for measuring and analysing the study outcomes will be aware of the treatment given.
  Study team will document consent to participate and non-objection response to classroom lighting change. A 100% non-objection rate from the parents of students within one classroom will be required prior to changing the classroom lighting. Randomization: Classrooms randomly be assigned into technical or other arms (cluster). Students from classrooms not included in the technical arms will be randomized into control or digital intervention arm.
  For the purpose of maintaining double-blind, all participants (parents) will be given LightUP application that will either be sham or interventional. Only a group of unmasked study personnel will know the treatment allocation and they will not be involved in data collection and analysis of results/data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Technical Intervention (n=132) (Experimental): Technical refinement of classroom lighting + Sham LightUP phone application (s-LightUP)
  Interventions: Other: Light Intervention
- Digital Intervention (n=132) (Experimental): Standard classroom lighting + Interventional LightUP phone application (i-LightUP)
  Interventions: Behavioral: Digital Intervention
- Control Group (n=132) (Placebo Comparator): Standard care or control group which involves standard classroom lighting + Sham LightUP app (s-LightUP).
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Light Intervention — LEDs mimicking the spectrum of sunlight (4000K) administered daily for 1 academic year, every school day, for the entire school day. The light levels generated by these LEDs will fluctuate throughout the day but will remain under 1000 lux.
  Arms: Technical Intervention (n=132)
Behavioral: Digital Intervention — Smart-phone application (LightUP) will be synced daily to a child-worn light and activity sensor and will allow parents to track their children's outdoor time and exposure to brighter light levels across the day. The application will also nudge parents to increase their child's exposure to light (e.g., increase time outdoors, or sitting next to a window indoors) after school hours for better myopia prevention and control. i-LightUP aims to gradually assist parents in helping their children reach the ultimate goal of spending at least 2 hours per day in brighter light conditions (e.g., above 1000 lux).
  Arms: Digital Intervention (n=132)
Other: Control Group — Standard Classroom Lighting + Sham LightUP phone application
  Arms: Control Group (n=132)

SUMMARY:
The goal of this clinical trial is to evaluate whether the optimization of daily exposure to light in primary school children can lead to better myopia prevention and control. The trial also aims to better understand the impact of light exposure on sleep and cognitive performance in children.

This trial has 3 arms namely, (1) a technical intervention arm, (2) a digital intervention arm, and (3) a control arm.

1. technical intervention - which involves changing of classroom lighting in primary schools to ceiling lights that mimic the spectral composition of sunlight and fluctuates in intensity. Parents of children within that arm will have a sham smart-phone application (s-LightUP)
2. digital intervention - which involves standard classroom lighting and giving parents an interventional smart-phone application (i-LightUP) that will be coupled with their child's light and activity sensor (wrist worn device ). The interventional app will provide individually tailored recommendation based on their children's behaviour (data feedback that is collected from the light and activity monitoring watch). The interventional app would then send reminder prompts/notifications to encourage parents help their children achieve required amounts of myopia-preventive light quantum target set per day.
3. Standard care or control group which involves standard classroom lighting and parents having a sham smart-phone application (s-LightUP)

Participants will:

* be randomised to receive either no intervention (control group), technical intervention (light intervention that mimics sunlight) or digital intervention (parents having an app that syncs with child's light and activity sensor which will provide feedback to parents to encourage and recommends increment of outdoor activities and hours).
* have their myopia progression monitored every 6 monthly and cognitive assessment done once every 3 months over a year.
* wear the light and activity sensor watches throughout the 1-year study period as much as possible (minimum 1 week per month) except for wet water activities such as swimming, diving and showering for research data collection purpose.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate whether the optimization of daily exposure to light in primary school children can lead to better myopia prevention and control. To do so, we will evaluate the effectiveness, safety and feasibility of:

1. Arm 1: technical intervention which involves spectro-temporal refinement of classroom lighting in primary schools using full spectrum light emitting diodes (LEDs) (CCT: 4000K) in addition to intermittent fluctuations in light levels. Parents of children in that arm will have access to a sham version of the LightUP mobile application to facilitate communication with the study team and questionnaire collection during the study.
2. Arm 2: digital intervention which involves optimization of daily light exposure using an individualised behaviour-changing smart-phone application (Interventional LightUP application) coupled with child-worn light and activity sensors to provide parents with an individually tailored recommendation to adapt their children's behaviour and provide them with the required amounts of myopia-preventive light quantum/day. + standard classroom lighting

   As compared to:
3. Arm 3: Standard care or control group which involves standard classroom lighting and no access to the interventional version of the LightUP application. Parents of children in that arm will have access to a sham version of the LightUP mobile application to facilitate communication with the study team and questionnaire collection during the study.

Our study will also lead to the following scalable and implementable outcomes:

1. evidence-based lighting designs and policy recommendations for classrooms;
2. a user-friendly, smart digital eyecare companion that aligns perfectly with Singapore's Smart Nation Initiative.

A secondary objective of this study is to better understand the impact of light exposure on sleep and cognitive performance in children. This will be achieved through continuous wrist actigraphy monitoring and through cognitive assessments, performed in classrooms, using tablets (one tablet/child). The assessment consists of validated, child-adapted, higher cognitive tasks testing the following constructs: impulse control, spatial working memory, content working memory, cognitive flexibility, reaction time, and processing speed.

ELIGIBILITY:
Inclusion Criteria:

* Subject must meet all the inclusion criteria below to participate in this study.

  1. Written Informed Consent form from parent / legal guardian and assent from child subject has been obtained
  2. Is between 7 to 10 years of age at start of study intervention which is 2 January 2025 or 1 January 2026
  3. Studying in either Primary 2 or 3 classes of the participating school(s) in academic year 2025 or 2026.
  4. Presenting visual acuity or best corrected visual acuity (BCVA) better or equal to LogMAR 0.2 (equivalent to Snellen 6/9 or better) in each eye
  5. Normal Intraocular pressure (not more than 21mmHg)
  6. No ocular conditions (e.g., optic nerve disease, glaucoma, retinal diseases) except for refractive error.
  7. No ocular conditions affecting the accuracy of the ophthalmic examinations
  8. In good general health with no significant systemic diseases that may affect eye health

     Exclusion Criteria:
* All subjects meeting any of the exclusion criteria at baseline will be excluded from participation.

  1. Previous or ongoing myopia control treatment (including but not limited to orthokeratology, atropine, pirenzepine, myopia control spectacle and contact lenses, light therapy)
  2. Ongoing participation in other myopia prevention and control research trials
  3. Any systemic or neurologic diseases (e.g. cancer, epilepsy, Kawasaki disease) known to affect eye health or make the participant vulnerable to the ophthalmic examinations (e.g., light flash)
  4. Any other conditions precluding adherence to the protocol including unwillingness to refrain from myopia control treatment for the duration of the study

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 396 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-01-26 (Estimated); Study Completion 2027-01-26 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic auto-refraction | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using autoref/kerato/pachy/tonometer
Axial Length | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using non-contact optical biometer
Choroidal Thickness | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using optical coherence tomography (OCT) scan

SECONDARY OUTCOMES:
Retinal and choroidal perfusion | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using optical coherence tomography angiography (OCT-A) function within OCT machine used to measure choroidal thickness.
Corneal Curvature | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using autoref/kerato/pachy/tonometer.
Corneal Thickness | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  Measured using autoref/kerato/pachy/tonometer.
Impulse control | 1 year, once every 3 months (Baseline, Month 3, Month 6, Month 9 , Month 12 Visit)
  Impulse control will be assessed using a validated, child-adapted task developed by collaborator Dr. Evelyn Law (NUS). The "Day and Night Cards" task or a similar task will be administered on tablets (one tablet per child). Impulse control will be quantified by the number of errors committed by the children during the task which involves shifting instructions and paradigms.
Cognitive flexibility | 1 year, once every 3 months (Baseline, Month 3, Month 6, Month 9 , Month 12 Visit)
  Cognitive flexibility will be assessed using a validated, child-adapted task developed by collaborator Dr. Evelyn Law (NUS). The "Day and Night Cards" task or a similar task will be administered on tablets (one tablet per child). Cognitive flexibility will be quantified by the number of errors committed by the children during the task which involves shifting instructions and paradigms.
Spatial working memory | 1 year, once every 3 months (Baseline, Month 3, Month 6, Month 9 , Month 12 Visit)
  Spatial working memory will be assessed using a validated, child-adapted task developed by collaborator Dr. Evelyn Law (NUS). The "Eight Boxes" task or a similar task will be administered on tablets (one tablet per child). Spatial working memory will be quantified by the number of errors committed by the children during the task.
Content working memory | 1 year, once every 3 months (Baseline, Month 3, Month 6, Month 9 , Month 12 Visit)
  Content working memory will also be assessed using a validated, child-adapted task developed by collaborator Dr. Evelyn Law (NUS). The "Eight Boxes" task or a similar task will be administered on tablets (one tablet per child). Content working memory will be quantified by the number of errors committed by the children during the task when remembering the content of different items in the task (e.g., strawberry, watermelon, etc.).
Processing speed | 1 year, once every 3 months (Baseline, Month 3, Month 6, Month 9 , Month 12 Visit)
  Processing speed will be assessed from the previous cognitive tasks (e.g., Eight Boxes and Day and Night Cards" through the investigation of reaction time (ms) in response to the content of the tasks. The tasks will be administered on tablets (one tablet per child).
Sleep quantity | 1 year or at least 1 week per month for 1 year
  This is a secondary outcome and will depend on the days of wear of the activity and light trackers. Night time sleep quantity (minutes) will be collected through actigraphy watches given to participants.
Sleep efficiency | 1 year or at least 1 week per month for 1 year
  This is a secondary outcome and will depend on the days of wear of the activity and light trackers. Night time sleep efficiency (%) calculated as the amount of time spent asleep (in minutes) by the total amount of time in bed (in minutes) will be measured using actigraphy watches given to participants.
Height | 1 year, at baseline and 12 months from baseline
  Height of the participant in cm
Weight | 1 year, at baseline and 12 months from baseline
  Weight of the participant in Kg
Visual acuity | 1 year, once every 6 months (Baseline, Month 6, Month 12 Visit)
  LogMAR visual acuity test

OTHER OUTCOMES:
Daytime average light levels (lux) | 1 year or at least 1 week per month for 1 year
  Daytime average light levels (lux) collected using wearable light sensors.
Daytime average melanopic lux | 1 year or at least 1 week per month for 1 year
  Daytime average melanopic lux collected using wearable light sensors.
Time spent outdoors (questionnaires) | 1 year or at least 1 week per month for 1 year
  Estimated time spent outdoors collected using questionnaires
Time spent outdoors (wearables) | 1 year or at least 1 week per month for 1 year
  Calculated time spent outdoors collected using the wearable light sensors.
Color vision | Baseline
  Color vision assessment using the Ishihara color vision test
Cover test (distance and near) | 1 year, repeated every 6 months
  Cover test to screen for strabismus

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P. Najjar, PhD, Principal Investigator — National University of Singapore
Locations (5):
- Singapore (5):
  - National University of Singapore, Yong Loo Lin School of Medicine, Department of Ophthalmology, Eye N Brain Research Lab, Singapore
  - Marymount Convent School, Singapore
  - Bedok Green Primary School, Singapore
  - Westwood Primary School, Singapore
  - Wellington Primary School, Singapore

IPD SHARING:
Plan to Share IPD: No